CLINICAL TRIAL: NCT05962736
Title: The Effect of Mirror Therapy on Shoulder Pain and Function in Patients Undergoing Thoracotomy
Brief Title: The Effect of Mirror Therapy After Thoracotomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Neriman Temel Aksu, Research Assistant (Expert Physiotherapist), Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: AkdenızUnıvesıty
Record Dates: First submitted 2023-07-19; First posted 2023-07-27 (Actual); Last update posted 2024-08-26 (Actual); Status verified 2024-08

CONDITIONS: Post-thoracotomy Pain Syndrome; Shoulder Pain
MeSH Terms: conditions — Shoulder Pain | interventions — Mirror Movement Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (No Intervention): The control group consisted of patients who underwent thoracotomy and underwent routine rehabilitation in the post-surgical period. routine respiratory rehabilitation program; It consists of a) positioning, b) general body exercises, c) airway clearance techniques, d) breathing exercises, e) incentive spirometry and f) mobilization applications.
- Study group (Experimental): The study group consisted of patients who would receive mirror therapy in addition to the routine rehabilitation program described above and applied to the control group in the post-thoracotomy period.
  Interventions: Device: Mirror therapy

INTERVENTIONS:
Device: Mirror therapy — The patients received a total of 24 sessions of treatment for 8 weeks, 3 sessions a week, starting from the postoperative 1st day after thorakaotomy. Each treatment session lasts between 60 and 90 minutes.
  Arms: Study group

SUMMARY:
After thoracotomy, limitation in shoulder functions, ipsilateral shoulder pain, decrease in shoulder muscle strength and deterioration in quality of life occur. The exercise program applied after thoracotomy includes active range of motion exercises, postural correction activities, scapular strengthening exercises, and stretching of the chest and shoulder muscles. Mirror therapy can improve motor functions and reduce unilateral pain. This study aims to evaluate the effects of upper extremity exercises based on mirror therapy after thoracotomy on ipsilateral shoulder pain, shoulder joint range of motion, shoulder muscle strength, shoulder function, quality of life, movement and fear of re-injury. The patients were divided into 2 groups as "mirror therapy group" and "control group", by choosing a simple randomization so that they could not see what was written on their pre-prepared papers. Standard medical treatment, care and pulmonary rehabilitation program were applied to both groups. In addition to the routine rehabilitation program after thoracotomy, the study group received a total of 24 sessions of foal therapy, 3 sessions a week, for 8 weeks. Data were collected using the Personal Information Form including the demographic characteristics of the patients, Tampa Kinesiophobia Scale, Numerical Pain Rating Scale (NPRS), Shoulder Active Range of Motion, Pain Catastrophization Scale, Shoulder Pain and Disability Index, Shoulder muscle strength, SF-12. performed before and after treatment.

DETAILED DESCRIPTION:
Pelvic examination has been a worrisome examination for women since the first years of gynecology science until today. Previous studies have discussed patient anxieties experienced during interventions such as radiological imaging, endoscopy, colonoscopy, bronchoscopy, and invasive cardiac interventions. Short informative videos that do not cause any cost loss or harm increase the tolerance with these applications and reduce patient anxiety. Additionally, many studies have emphasized that doctors have no time to provide information trainings for the vaginal examination among their intense practices. Information that cannot be provided before the gynecologic examination due to limited time causes pelvic pain in women due to the anxiety experienced during the examination. In the literature, the concept of chronic pelvic pain is defined as non-cyclical pain that lasts longer than six months and develops the area below the umbilicus and between the gluteal lines; however, pelvic pain is observed depending on the excessive activity of pelvic floor muscles during the examination in patients who have the fear of the gynecologic examination.

The aim of this study is to evaluate the effect of multimedia patient information training provided before the gynecologic examination on the patient's pelvic pain, anxiety, and fear.

The present study is designed as a randomized controlled single-blind prospective experimental study to examine the effects of patient training provided before the gynecologic examination on the patient's anxiety, fear, and pelvic pain.

The study is conducted with 80 voluntary patients in the age range of 18-50 years, who applied to the gynecology and obstetrics clinic.

The inclusion criteria are as follows; having no known cerebrovascular disease, having no morbid obesity and heart disease that would pose an obstacle to the study, having no cognitive disorder that would pose an obstacle to communication, having no stroke and the associated influence, and agreeing to participate in the study.

Participants are grouped as; who were gived information about vaginal examination in the training group (n=40) and who are not gived information about vaginal examination in the control group (n=40) groups. Randomization is performed by using the sealed envelope method, just before the evaluations. Vaginal examination information is video based patient education programme. That contained pelvic anatomy and how to practice vaginal examination by gynecologists.

Age, weight and height measurements, educational background, occupation, marital status, gravidity and parity, number of gynecologic examinations, presence of dyspareunia and dysmenorrhea, urinary incontinence complaints, smoking and alcohol habits of the patients in both groups are recorded. Clinical evaluation is carried out to provide information about the patients' demographic characteristics and medical condition. The patient completed the questionnaires. The researcher helped patients who does not understand the questions.

Primary result measurements are performed using the State-Trait Anxiety Inventory (STAI-1-2) and the Visual Analog Scale (VAS). Anxiety level is evaluated using the STAI-1,2; whereas, pelvic pain, anxiety and pain level are assessed using the VAS.

STAI-2 is applied only once after obtaining personal information in the beginning of the study. All other measurements are repeated three times as before the training, after the training and after the examination for the control group. The measurements are repeated twice as before the examination and after the examination for the control group.

All the individuals in the training group watch a short video about the examination procedure before the examination and are given training via multimedia information. The training consist of a 5-minute video about the detailed examination procedure. The individuals in the control group are not given the training.

The data are analyzed in the SPSS 18.0 (Statistical Package for Social Sciences) program. Descriptive statistical methods were chosen for demographic data. The chi-square test is used for the comparison of demographic rates between the groups and the Fisher's exact test is used if the expected frequencies are not met. Significance of the difference between the groups in terms of mean values is evaluated using the Student's t test. In cases in which parametric test assumptions are not met, the Mann Whitney-U test or the Wilcoxon test, which are non-parametric counterparts of these tests, is used. In all the tests, the value of p<0.05 is accepted to be statistically significant.

While conducting the study, scientific principles and universal ethical principles is followed. Accordingly, the study is conducted based on principles of informed consent, autonomy, confidentiality and protection of privacy, justice, and nonmaleficence/beneficence. As the use of human phenomenon requires the protection of individual rights in studies, the Declaration of Helsinki on Human Rights is followed throughout the study. In order to conduct the study; written permissions are obtained from Akdeniz University Hospital Department of Obstetrics and Gynecology, and from Akdeniz University Clinical Research Ethics Committee before starting the study.

ELIGIBILITY:
Inclusion Criteria:

* Patients who were hospitalized in Akdeniz University Hospital Thoracic Surgery Clinic and underwent lung resection with standard posterolateral thoracotomy (lobectomy, segmentectomy or wedge resection),
* Those between the ages of 25-65,
* Hemodynamically stable,
* Those who were extubated at the 2nd or 3rd postoperative hour and who did not develop any complications after extubation,
* No known cerebrovascular disease,
* Not having morbid obesity and heart disease that will prevent working,
* Does not have cognitive and cognitive impairments that will prevent communication,
* No previous paralysis and related effects,
* Individuals who agree to participate in the study.

Exclusion Criteria:

* Those who stayed in the intensive care unit for more than 4 days in the postoperative period,
* Those who have had another surgical procedure within 6 months,
* Those with postoperative cooperation problems such as delirium,
* Those with Rotator Cuff injuries,
* Those with cervical radiculopathy,
* Those with rheumatological diseases,
* Those with neurological disease,
* Those with a history of dislocation, subluxation,
* Those with a history of fracture,
* Those with congenital deformity,
* Those who have a history of surgery related to the shoulder,
* Those who have trouble perceiving tests and exercises

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 70 (Actual)
Dates: Start 2022-03-06 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-07-12 (Actual)

PRIMARY OUTCOMES:
Change of Pain Score | Change from Baseline Pain Score at 8 weeks.
  Numerical Pain Rating Scale (NPRS) was used as a one-dimensional scale for pain
Change of Active Shoulder Range of Motion | Change from Baseline Active Shoulder Range of Motion at 8 weeks.
  Active shoulder range of motion of the patients will be evaluated with a digital goniometer (Baseline Digital Absolute & Axis Goniometer) using a standard protocol. Total shoulder motion that allows motion of all joints in the shoulder complex will be measured, glenohumeral motion will not be isolated. Flexion, abduction, external and internal rotation of the shoulder will be evaluated. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Shoulder Muscle Strength | Change from Baseline Shoulder Muscle Strength at 8 weeks.
  Shoulder muscle strength will be measured using a dynamometer (MicroFET 2 Manual Muscle Tester). Force measurements will be taken for shoulder flexion, abduction, internal and external rotation. Before starting the test, patients will be informed about how to perform the test. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated.
Change of Quality of Life Score | Change from Baseline Quality of Life Score at 8 weeks.
  The quality of life of our patients will be evaluated using the Short Form-12. Health-related
Change of Shoulder, Pain and Disability Index Score | Change from Baseline Shoulder, Pain and Disability Index Score at 8 weeks.
  Shoulder function will be measured using the Shoulder, Pain and Disability Index , a self-rated questionnaire designed to measure shoulder pain and disability. Shoulder Pain and Disability Index is a reliable questionnaire evaluating shoulder pain and disability. Turkish reliability and validity were performed by Bumin et al. in 2008. There are 2 subscales and 13 items in total in the index. 5 of them evaluate pain and 8 evaluate disability. The items of both subscales are measured with a visual analog scale from 0 to 10. The scores given by the individual are added together and calculated as a percentage. Higher scores indicate more severe pain and higher disability. Preoperative period, postoperative 7th day, postoperative 4th week and postoperative 8th week will be repeated
Change of Tampa Kinesiophobia Scale | Change from Baseline Tampa Kinesiophobia Scale Score at 8 weeks.
  This scale, which is frequently used in the literature, is based on avoidance due to fear, fear in work-related activities, fear of movement or re-injury. Tampa Kinesiophobia Scale is a 17-item scale developed to measure fear of movement and re-injury. The scale includes parameters of injury/re-injury and fear-avoidance in work-related activities. The fact that it is an important outcome parameter for physiotherapists in evaluating the success of the treatment and especially the social participation of the patients, and being a scale that can be used in various patient groups, makes Tampa Kinesiophobia Scale a valuable measurement parameter in the clinic. Tampa Kinesiophobia Scale is a 4-point Likert scale scored as 1-strongly disagree, 2-disagree, 3-agree, 4-strongly agree. The total score is calculated after questions 4, 8, 12 and 16 are reverse scored one by one. The total score is between 17-68. A high value in Tampa Kinesiophobia Scale indicates a high level of kinesiophobia.

SECONDARY OUTCOMES:
Height in Meters | Initial assessment before surgery.
  The height of all subjects in meters (m) will be noted before the surgery.
Weight in Kilograms | Initial assessment before surgery.
  The weight of all subjects in kilograms (kg) will be noted before the surgery.
Body Mass Index (BMI) in kg/m^2 | Initial assessment before surgery
  Body Mass Index (BMI) will be calculated with the formula weight (kg)/height (m)^2.

CONTACTS AND LOCATIONS:
Overall Officials: Neriman T Aksu, Principal Investigator — Akdeniz Üniversitesi Antalya Sağlık Yüksekokulu
Locations (1):
- Neriman Temel Aksu, Antalya, Turkey (Türkiye)

REFERENCES:
- [Derived] Aksu NT PhD, Baskurt Z, Keskin H. Effects of Mirror Therapy-Based Upper Extremity Exercises After Thoracotomy: A Randomized Controlled Trial. Pain Manag Nurs. 2025 Aug;26(4):e411-e420. doi: 10.1016/j.pmn.2025.02.003. Epub 2025 Mar 7. PMID 40057453